CLINICAL TRIAL: NCT03413306
Title: A Phase II Multicenter Randomized Study of Eltrombopag Combined With Cyclosporine and hATG Versus hATG and CsA as First Line Treatment in Pediatric Patients With Severe Acquired Aplastic Anemia
Brief Title: Eltrombopag+hATG+CsA vs. hATG+CsA in Children With Severe AA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2016-01
Record Dates: First submitted 2017-12-22; First posted 2018-01-29 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Acquired Aplastic Anemia
Keywords: aplastic anemia; immunosupressive therapy; ATG; eltrombopag
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eltrombopag + IST (ATG + CsA) (Experimental)
  Interventions: Drug: Eltrombopag; Drug: IST (ATG + CsA)
- IST (ATG + CsA) (Active Comparator)
  Interventions: Drug: IST (ATG + CsA)

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag is an oral mimetic thrombopoietin selectively binding transmembrane and juxtamembrane domains of the thrombopoietin receptor different from the binding site of thrombopoietin. Therefore it does not compete for binding with the native molecule. It is promoting thrombopoiesis and release platelets from mature megakaryocytes. Also it promotes more primitive multilineage progenitors and hematopoietic stem cells to proliferate and differentiate into thrombocytes, erythrocytes and leukocytes.
  Other Names: Revolade
  Arms: Eltrombopag + IST (ATG + CsA)
Drug: IST (ATG + CsA)
  Other Names: controle

SUMMARY:
The analysis of our own clinical data suggests that majority of the hematologic responses observed after the course of h-ATG/CsA is partial, and about 10% tend to have cyclosporine dependence.

The aim of the current study is to improve the rate and the quality of hematologic response as well as to prevent delayed complications such as relapse and clonal progression by means of adding eltrombopag to standard immunosuppressive therapy

DETAILED DESCRIPTION:
This trial will evaluate safety and efficacy of combination eltrombopag with standard hATG/CSA as first line therapy in patients with SAA. The primary endpoint is going to be estimating the rate of complete hematologic response at the point in four months after the end of the treatment. Secondary endpoints are probability of relapse, hematologic blood count recovery in 6 and 12 months after the treatment, survival, clonal evolution into myelodysplasia and leukemia

Aplastic anemia can be treated effectively with allogeneic bone marrow transplantation and immunosuppressive therapy with horse anti-thymocyte globulin (h-ATG) and cyclosporine (CsA), allowing to achieve a comparable long-term survival about 80%. However, one third of the patients treated with h-ATG/CsA, does not respond, and 25-30% of the responders relapse. The analysis of our clinical data suggests that majority of the hematologic responses observed following initial h-ATG/CsA are partial, with only a few patients achieving normal blood counts, and about 10% tend to have cyclosporine dependence. Although horse ATG/CsA provides represented a major advance in the treatment of SAA, such condition as refractory course of the disease, incomplete response, relapse, and clonal evolution limit the success of this treatment. Thus, new regimens are needed to overcome these limitations and provide a better alternative to stem cell transplantation.

One option of improving the quality of hematologic responses is influencing underlying stem cell function. Previous attempts to improve response by hematopoietic cytokines, including erythropoietin and G-CSF, have failed. Thrombopoietin is the principal endogenous regulator of platelet production. In addition, TPO also has stimulatory effects onto primitive multilineage progenitors and stem cells in vitro and animal models. Eltrombopag (Revolade), an oral 2nd generation small molecule TPO-agonist, is approved for treatment of chronic immune thrombocytopenic purpura and SAA who had insufficient response to immunosuppressive therapy. Eltrombopag increases platelets in healthy subjects and in thrombocytopenic patients, and recently has showed clinically significant hematologic responses in refractory SAA patients. The aim of this tudy to improve hematologic response rate and its quality, as well as to prevent late complications such as relapse and clonal progression, by adding eltrombopag into standard immunosuppressive therapy This trial evaluates safety and efficacy of combining eltrombopag with standard hATG/CSA as the first line of therapy in patients with SAA. The primary endpoint is going to be estimation of the rate of complete hematologic response in 4 months. Secondary endpoints are probability of relapse, robust hematologic blood count recovery in 6 and 12 months after the treatment, survival, clonal evolution to myelodysplasia and leukemia.

This is a trial aiming to increase 4 months overall response rate. The sample size is calculated on the hypothesis that the experimental treatment will increase the 4 months response rate in 20% in comparison with standard IST treatment arm. Under these assumptions, the sample size to reject the null hypothesis is n=100 patients, 50 patients in each treatment arm; alpha-error 0.05; power 0.75.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of severe and very severe Aplastic anemia
2. 2 - 18 years old
3. Written informed consent signed by a parent or legal guardian prior to initiation of any study specific procedure.
4. Absence of HLA-identical family member

Exclusion Criteria:

1. myelodysplastic syndrome 4. Prior immunosuppressive therapy 5. Patients with hepatic, renal or cardiac failure, or any other life- threatening concurrent disease 6. hypersensitivity to any of the component medications 7. Creatinine >2.5 mg/dL× the upper limit of normal, 8. Total bilirubin >1.5 × the upper limit of normal mg/dL , 9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3-5 × the upper limit of normal

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12-10 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
ORR (CR + PR) | 4 months
  The primary objective of this trial is to investigate whether Eltrombopag added to standard immunosupressive treatment hATG and CsA increases the overal (partial + complete) response rate at four months in untreated children with severe aquired aplastic anemia.

SECONDARY OUTCOMES:
Platelet count | 4 and 6 months
Hemoglobin | 4 and 6 months
Neutrophil count | 4 and 6 months
Cumulative incidence of response | 4 and 6 months
Duration of hematologic response | 2 years
  Time from the date of the start of response to the date of relapse defined as again meeting criteria for severe or moderate aplastic anemia
Overall survival | 2 years
Event-free survival | 2 years
Cumulative incidence of relapse | 2 years
Cumulative incidences of clonal evolution | 2 years
Cumulative incidence of PNH population occurrence and clinical hemolytic PNH occurrence | 2 years
Cumulative incidence of adverce effects | 4 months
  Number of participants with severe adverse events (3-5 stage CTCAE v.4.0) associated with assessment of eltrombopag usage in patients with severe aplastic anemia in 4 months after first day of treatment. Death before evidence of adverce event is competing event.
Cumulative incidence of adverce effects | 4 months
  Number of participants with severe adverse events (3-5 stage CTCAE v.4.0) associated with assessment of eltrombopag dose in patients with severe aplastic anemia in 4 months after first day of treatment. Death before evidence of adverce event is competing event.
Comparison of cumulative incidence of adverce effects in two arms | 2 years
  comparison between two arms of number of participants with severe adverse events (3-5 stage CTCAE v.4.0) associated with treatment in patients with severe aplastic anemia in 2 years after first day of treatment with death before evidence of adverce event as a competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Galina Novichkova, Principal Investigator — Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology; Alexei Maschan, Principal Investigator — Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

REFERENCES:
- [Derived] Goronkova O, Novichkova G, Salimova T, Kalinina I, Baidildina D, Petrova U, Antonova K, Sadovskaya M, Suntsova E, Evseev D, Matveev V, Venyov D, Khachatryan L, Litvinov D, Pshonkin A, Ovsyannikova G, Kotskaya N, Gobadze D, Olshanskaya Y, Popov A, Raykina E, Mironenko O, Voronin K, Purbueva B, Boichenko E, Dinikina Y, Guseynova E, Sherstnev D, Kalinina E, Mezentsev S, Streneva O, Yudina N, Plaksina O, Erega E, Maschan M, Maschan A. Efficacy of combined immunosuppression with or without eltrombopag in children with newly diagnosed aplastic anemia. Blood Adv. 2023 Mar 28;7(6):953-962. doi: 10.1182/bloodadvances.2021006716. PMID 35446936